CLINICAL TRIAL: NCT00233844
Title: Studying the Analgesic Mechanism of the "Cough-Trick" - Randomized Crossover Volunteer Study
Brief Title: Studying the Analgesic Mechanism of the "Cough-Trick"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: III UV 82/03
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2005-10-06 (Estimated); Status verified 2005-10

CONDITIONS: Pain; Acute Pain; Venipuncture
Keywords: Acute pain; pain on venipuncture; "cough-trick"; distraction
MeSH Terms: conditions — Pain; Acute Pain | interventions — Phlebotomy

INTERVENTIONS:
Procedure: Venipuncture with "cough-trick"

SUMMARY:
The aim of the trial is to study the possible mechanism of the pain reducing effect of CT at peripheral venipuncture

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers aged 20-40 years, height 165-190 cm.
2. Physical status I according to American Society of Anesthesiologists (ASA) classification.
3. Straight run of the vein on the dorsum of the non-dominant hand at least 4 cm long and 3 mm thick
4. No analgesics, anticoagulants and/or antiplatelet agents, sedatives or alcohol

Exclusion Criteria:

1. History of peripheral neuropathy
2. Abnormal skin conditions (infection, scars, psoriasis, eczema)
3. Unsuccessful venipuncture
4. Inflamed site of VP within 1 week after VP

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21
Dates: Start 2004-02

PRIMARY OUTCOMES:
Pain intensity measured on VAS-100 scale

SECONDARY OUTCOMES:
Heart rate, arterial pressure, hand withdrawal, sweating

CONTACTS AND LOCATIONS:
Overall Officials: Taras I. Usichenko, Assistant Professor, Principal Investigator — Anesthesiology and Intensive Care Medicine Department, Ernst Moritz Arndt University of Greifswald, Germany